CLINICAL TRIAL: NCT05405179
Title: Simultaneous Dental Implant in Free Vascularized Bone Flaps for Jaw Reconstruction Using Patient-specific Surgical Guides and Titanium Plates: a Pilot Study
Brief Title: Simultaneous Dental Implant in Free Vascularized Bone Flaps for Jaw Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW21-341
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-05

CONDITIONS: Mandibular Reconstruction; Dental Implant; Free Tissue Flaps; Jaw Neoplasms
Keywords: Maxillo-mandibular reconstruction; jaw neoplasms; free tissue flaps; dental implant; Patient-specific titanium plates; virtual surgical planning
MeSH Terms: conditions — Jaw Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simultaneous dental implantation (Experimental): To perform dental implantation simultaneously in free vascularized flap during jaw reconstruction
  Interventions: Procedure: Simultaneous dental implantation

INTERVENTIONS:
Procedure: Simultaneous dental implantation — To perform dental implantation simultaneously in free vascularized bone flaps for jaw reconstruction using patient-specific surgical guides and titanium plates

SUMMARY:
After jaw resection, free vascularized bone flaps are frequently used for repairing maxillofacial defects. Simultaneous dental implantation is more preferable to secondary implantation as it saves the patients from going through a second surgery after recovering from the first one.

In this study, the aim is to preliminarily evaluate the clinical outcome of simultaneous dental implants in vascularized bone flaps in jaw reconstruction using patient-specific surgical plates and 3-in-1-PSSG. The objectives of this study were: 1) to investigate the intraoperative success rate; 2) to measure the accuracy of dental implants position; and 3) to assess implant survival rate and postoperative adverse events.

DETAILED DESCRIPTION:
After jaw resection, free vascularized bone flaps are frequently used for repairing maxillofacial defects. Owing to the extensive loss of dentition and soft tissues after the ablative surgery, the use of conventional fixed and removable prostheses is often limited in such cases. Implant-supported fixed prosthesis could be a better alternative which is free-standing and does not rely on tooth or soft tissue support. Dental implants on bone flaps restore the patient's oral function and comfort. Simultaneous dental implantation is more preferable to secondary implantation as it saves the patients from going through a second surgery after recovering from the first one.

However, conventional freehand immediate placement of dental implants in jaw reconstructive surgery is technically challenging as the position has to be highly precise to support an aesthetic and functional prosthesis. The current development of computer-aided surgery has been able to plan the inset of a vascularized bone flap in the maxillomandibular complex using digitally planned and printed surgical guides based on the patient's computed tomography (CT) data. The computer-aided surgery also facilitates the placement of dental implants at the optimal position and the modification of the bony reconstruction according to the implant position. Previously, the investigators have designed and fabricated novel patient-specific surgical plates by metal three- dimensional (3D) printing technology for jaw reconstruction, which led to precise reconstructive outcomes. In this study, the investigators propose a novel three-in-one patient-specific surgical guide (3-in-1-PSSG) which includes bone segmentation, surgical plate and implant placement positioning functions, to facilitate simultaneous dental implants in vascularized bone flap jaw reconstruction. It is hypothesized that the 3-in-1-PSSG simplifies the surgical procedure. Together with the patient-specific titanium plate, the clinical outcomes for simultaneous dental implants in jaw reconstruction with vascularized bone flap will be improved.

In this study, the aim is to preliminarily evaluate the clinical outcome of simultaneous dental implants in vascularized bone flaps in jaw reconstruction using patient-specific surgical plates and 3-in-1-PSSG. The objectives of this study were: 1) to investigate the intraoperative success rate; 2) to measure the accuracy of dental implants position; and 3) to assess implant survival rate and postoperative adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years, of both gender;
2. Diagnosed with maxillofacial benign or malignant pathology and indicated for jaw surgery with immediate dental implants;
3. Titanium plates and dental implants will be used in the surgery;
4. Agree to comply with follow-up procedures;
5. Provision of signed and dated informed consent form.

Exclusion Criteria:

1. Patients who are pregnant;
2. Patients who need jaw reconstruction for the management of post-traumatic, congenital or developmental jaw deformities;
3. Patients who have medically compromised conditions and cannot tolerate the surgery;
4. Patients who are unable to have a two-week period prior to surgery, for virtual surgery simulation, patient-specific plates designing and fabrication;
5. Patients whose systemic conditions or diseases that violate the normal bone healing;
6. Patients who are unable to take the preoperative and postoperative CT/CBCT scans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative success rate | Intraoperative
  Success is defined as the uneventful placement of dental implant with adequate stability and correct angulation (Implant insertion torque value greater than 15Ncm and no implant thread exposure)

SECONDARY OUTCOMES:
Accuracy of dental implant placements | One month after surgery
  Position of dental implant on CT scan compared to planned position
Implant survival | 6 months after surgery
  Implant that is retained in the reconstructed jaw at the time of examination, regardless of the state of the prosthesis. or patient satisfaction.
Impact of oral health condition on quality of life | 6 months after surgery
  OHIP-14 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Philip Dental Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No